CLINICAL TRIAL: NCT02996149
Title: Endoscopic Lung Volume Reduction Coil Treatment in Patients With Chronic Hypercapnic Respiratory Failure
Status: Terminated | Type: Observational
Why Stopped: Technique no longer available
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Hans Klose, Dr., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV-5379
Record Dates: First submitted 2016-11-16; First posted 2016-12-19 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Endoscopic lung volume reduction coil treatment

SUMMARY:
Endoscopic lung volume reduction coil treatment is a treatment option for selected patients with severe emphysema. In the advanced stages, emphysema may lead to chronic hypercapnic respiratory failure. In this observational study the safety and efficacy of endoscopic lung volume reduction coil treatment in patients with chronic hypercapnic respiratory failure is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with emphysema (chronic obstructive pulmonary disease with forced expired volume in one second (FEV1) < 50% predicted and residual volume (RV) ≥ 200% predicted) in whom endoscopic lung volume reduction coil treatment is performed
* Chronic hypercapnic respiratory failure (PaCO2 ≥ 50 mmHg)
* Informed consent

Exclusion Criteria:

* Therapeutic anticoagulation
* Anti-platelet therapy exceeding the use of acetylsalicylic acid
* Severe pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe emphysema and chronic hypercapnic respiratory failure, in whom endoscopic lung volume reduction coil treatment is performed
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in PaCO2 | 3 months after endoscopic lung volume reduction (ELVR)

SECONDARY OUTCOMES:
Changes in PaCO2 | 6 and 12 months after ELVR
Changes in FEV1 | 3, 6 and 12 months after ELVR
Changes in vital capacity | 3, 6 and 12 months after ELVR
Changes in residual volume | 3, 6 and 12 months after ELVR
Changes in 6-minute walk distance | 3, 6 and 12 months after ELVR
Changes in quality of life (St. George's Respiratory Questionnaire, SGRQ) | 3, 6 and 12 months after ELVR
Changes in BMI | 3, 6 and 12 months after ELVR

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany